CLINICAL TRIAL: NCT05988892
Title: Improving Physical Activity in Rural Cancer Survivors
Brief Title: A Study of Physical Activity in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-001462; NCI-2023-05387 (Other: Clinical Trials Reporting Program)
Record Dates: First submitted 2023-07-26; First posted 2023-08-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
Keywords: Rural; Physical Activity
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Community Oncology patients entering cancer survivorship (Experimental): Patients participate in a virtual cancer rehabilitation program with weekly virtual visits by a cancer exercise specialist who provides a personalized synchronous exercise plan and receive bi-weekly phone calls/emails over 12 weeks. Patents also wear a Fitbit on study.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Use Exercise to increase physical activity (PA), as measured by cardiovascular endurance, muscular strength, and balance in underserved cancer survivors >60 years of age and/or those of any age residing at a rural address and to increase quality of life (QOL), as measured by physical functioning and fatigue, in underserved cancer survivors >60 years of age and/or those of any age residing at a rural address.

SUMMARY:
The purpose of this study is to determine if increasing physical activity (PA) will increase physical functioning, as measured by cardiovascular endurance, muscular strength, and balance in underserved adult cancer survivors > 60 years of age and/or those of any age residing at a rural address. Also, to determine if increasing PA will increase quality of life (QOL), as measured by physical functioning and fatigue, in underserved cancer survivors >60 years of age and/or those of any age residing at a rural address.

ELIGIBILITY:
Inclusion Criteria:

* Adult, cancer survivors (no active disease) at Mayo Clinic Health System (MCHS) in Northwest Wisconsin (NWWI), Southwest Wisconsin (SWWI), Southeast Minnesota (SEMN), or Southwest Minnesota (SWMN)
* Any stage cancer
* Age ≥18 years residing at a rural address (as defined by Rural America, census.gov)
* Completed active treatment of surgery, (neo)adjuvant chemotherapy, and/or (neo) adjuvant radiation. Patients receiving adjuvant endocrine therapy, targeted therapy, or immunotherapy therapies are eligible.
* Ownership of a computer/tablet/smartphone with internet access.
* Willingness to create a google account and maintain the account for use of the Fitbit
* Willingness and ability to attend study visits.
* Must be able to complete semi-tandem (10 seconds), side-by-side tandem [10 seconds and short physical performance batters(SPPB)] Score of 6 or greater to qualify for virtual exercise.
* Must be ambulatory without the use of assisted device(s).

Exclusion Criteria:

* Receiving surgery, (neo)adjuvant chemotherapy, (neo) adjuvant radiation, palliative treatment
* Are already performing >150 minutes/week of moderate activity or 75 min/week of vigorous physical activity
* Cancer-free for greater than 5 years
* Unable to complete weekly interventions/exercise due to traveling or unable to be active for more than 7 consecutive days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Change in physical functioning using Short Physical Performance Battery | Baseline; 12 weeks
  Change in physical functioning based on improvement in endurance, strength, and balance assessed using Short Physical Performance Battery (SPPB) pre- and post-12-week exercise intervention.
Change in Quality of Life (QOL) using Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline; 12 weeks
  QOL evaluated based on physical functioning and fatigue, assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) pre- and post-12-week exercise intervention.
Change in satisfaction using a 5-point Likert scale | Baseline; 12 weeks
  Satisfaction assessed using a 5-point Likert scale following 12-week exercise intervention and participant-reporting likelihood of recommending program.
Rate of adherence to program based on participation in virtual exercise sessions | Baseline; 12 weeks
  Adherence evaluated based on participation in virtual exercise sessions during 12-week exercise intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kaye T. Sturz, APRN, CNP, Principal Investigator — Mayo Clinic Health System in Eau Claire
Locations (4):
- United States (4):
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System-Mankato, Mankato, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials